CLINICAL TRIAL: NCT03654157
Title: A Non-interventional Study to Estimate the Rates of Outcomes in ACS Patients in Moscow
Brief Title: ACS Registry - A Non-interventional Study to Estimate the Rates of Outcomes in ACS Patients in Moscow
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00279
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Heart Attack; Stroke; Cardiovascular Death
MeSH Terms: conditions — Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Cardiovascular diseases (CVD) are currently the leading cause of death in industrialized countries and are expected to become the leading cause of death in emerging countries by 20201. According to the official Russian statistics, in 2015, CVD was the cause in 34% of deaths in Russia2.

Acute Coronary Syndrome (ACS) is the most prevalent manifestation of CVD and is associated with high mortality and morbidity. No other life-threatening disease is as prevalent or expensive to society3. In 2014 in Russian Federation 46 250 people died from acute myocardial infarction (MI) and 17 605 people died from recurrent MI4.

ACS is a clinical syndrome characterized by unstable angina (UA), non-ST-segment elevation myocardial infarction (NSTEMI) and ST-segment elevation myocardial infarction (STEMI). The most common cause of ACS is reduced myocardial perfusion that results from coronary artery narrowing caused by the formation of partially or totally occlusive thrombi in response to rupture of atherosclerotic plaques on the vessel wall5-7.

In Russian Federation ACS management after ACS is provided in out-patient settings by doctors of different specialties (cardiologists and general practitioners (GPs)). However, the management of ACS in out-patient settings in some regions in Russian Federation is frequently suboptimal. Moscow city significantly differs from other parts of Russia from ACS management at hospital stage (up to 90% of PCI managed ST elevation myocardial infarction (MI) patients, no thrombolysis, short first medical contact to balloon time etc.) but it is unclear if management of post MI patients in Moscow out-patient settings is also optimal. In-hospital mortality in MI patients decreased last years but there is no data on clinical outcomes during 12 months after MI in Moscow.

This study will provide the epidemiological data about rates of major adverse cardiovascular and cerebrovascular events (MACCE) (MI, stroke, cardiovascular death) within 12 months after MI in real clinical practice in Moscow and describe DAPT at out-patient setting. The information received in this study will help to optimize management of Russian patients with ACS. The data will be used in discussion with payers

ELIGIBILITY:
Inclusion Criteria:

The subject population that will be observed in this prospective study must meet the following criteria:

1. Patients survivors who visited outpatient setting after discharge from hospital due to MI (STEMI or NSTEMI) within 1 month after discharge from hospital;
2. Obtained written informed consent for participation in this study.
3. Age of 18 year or older.

Exclusion Criteria:

1. Current participation in a clinical study.
2. Unknown type of MI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who survived myocardial infarction and who come for further treatment and observation to polyclinic after discharge from hospital will be enrolled in this study if a patient provides a consent form. It is estimated that at least 2500 post MI patients are to be enrolled in the study. It is also assumed that the total size of the study population could be up to 10 000 post MI patients who are observed in polyclinics of Moscow city within first year after index event.
Sampling Method: Probability Sample
Enrollment: 1576 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
the cumulative incidence of Major Adverse Cardiovascular and Cerebrovascular Events (MACСE) | 1 year
  The primary objective of this study is to describe the cumulative incidence of Major Adverse Cardiovascular and Cerebrovascular Events (MACСE) [MI, stroke, and cardiovascular death] observed over 1 year after index MI in all patients enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Pesheva, Principal Investigator — GBUZ GP # 121 DZM; Tatyana Yurchak, Principal Investigator — GBUZ GP # 52 DZM; Veronika Vovk, Principal Investigator — GBUZ GP # 2 DZM; Dmitriy Privalov, Principal Investigator — GBUZ GKB # 51 DZM; Maria Klepikova, Principal Investigator — GBUZ GKB # 13 DZM; Olga Belkorey, Principal Investigator — GBUZ GP # 218 DZM; Natalya Karabinskaya, Principal Investigator — GBUZ GP # 19 DZM; Natalya Bosyakova, Principal Investigator — GBUZ GP # 19 DZM; Marina Lepatova, Principal Investigator — GBUZ GP # 107 DZM; Elena Dorofeeva, Principal Investigator — FGBU "Polyclinic # 1" Administrative Department of the President of the Russian Federation; Irina Shoshina, Principal Investigator — GBUZ GP # 109 DZM; Darya Semenova, Principal Investigator — GBUZ GP # 23 DZM; Elena Zherebetskaya, Principal Investigator — GBUZ KDC # 2 DZM; Marina Yarygina, Principal Investigator — GBUZ GP # 175 DZM; Elena Lukinskaya, Principal Investigator — GBUZ GP # 115 DZM; Irina Borovikova, Principal Investigator — GBUZ GP # 209 DZM; Tatiana Sladkova, Principal Investigator — GBUZ GP # 22 DZM; Elena Demyanova, Principal Investigator — GBUZ GP # 64 DZM
Locations (1):
- Research Site, Moscow, Moscow/Russia, Russia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Davies MJ. The pathophysiology of acute coronary syndromes. Heart. 2000 Mar;83(3):361-6. doi: 10.1136/heart.83.3.361. No abstract available. PMID 10677422
- [Background] Task Force for Diagnosis and Treatment of Non-ST-Segment Elevation Acute Coronary Syndromes of European Society of Cardiology; Bassand JP, Hamm CW, Ardissino D, Boersma E, Budaj A, Fernandez-Aviles F, Fox KA, Hasdai D, Ohman EM, Wallentin L, Wijns W. Guidelines for the diagnosis and treatment of non-ST-segment elevation acute coronary syndromes. Eur Heart J. 2007 Jul;28(13):1598-660. doi: 10.1093/eurheartj/ehm161. Epub 2007 Jun 14. No abstract available. PMID 17569677
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Alpert JS, Eagle KA, Faxon DP, Fuster V, Gardner TJ, Gregoratos G, Russell RO, Smith SC Jr. ACC/AHA guidelines for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on the Management of Patients With Unstable Angina). J Am Coll Cardiol. 2000 Sep;36(3):970-1062. doi: 10.1016/s0735-1097(00)00889-5. No abstract available. PMID 10987629
- [Background] Vasilyeva EY, Plavunov NF, Kalinskaya AI, Sapina AI, Vvedensky GA, Lebedeva AY, Skrypnyk DV, Shpektor AV. [Treatment of Patients With Acute Myocardial Infarction With ST-Segment Elevation. Organization of the Myocardial Infarction Network in Moscow]. Kardiologiia. 2016 Dec;56(12):48-53. No abstract available. Russian. PMID 28290804
- [Background] Jernberg T, Hasvold P, Henriksson M, Hjelm H, Thuresson M, Janzon M. Cardiovascular risk in post-myocardial infarction patients: nationwide real world data demonstrate the importance of a long-term perspective. Eur Heart J. 2015 May 14;36(19):1163-70. doi: 10.1093/eurheartj/ehu505. Epub 2015 Jan 13. PMID 25586123
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Hicks KA, Tcheng JE, Bozkurt B, Chaitman BR, Cutlip DE, Farb A, Fonarow GC, Jacobs JP, Jaff MR, Lichtman JH, Limacher MC, Mahaffey KW, Mehran R, Nissen SE, Smith EE, Targum SL. 2014 ACC/AHA Key Data Elements and Definitions for Cardiovascular Endpoint Events in Clinical Trials: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Data Standards (Writing Committee to Develop Cardiovascular Endpoints Data Standards). J Am Coll Cardiol. 2015 Jul 28;66(4):403-69. doi: 10.1016/j.jacc.2014.12.018. Epub 2014 Dec 29. No abstract available. PMID 25553722
- See also: CSR synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00279&attachmentIdentifier=e84544ce-905e-44fd-b84b-ef96ee81ac03&fileName=CSR_synopsis_redacted.pdf&versionIdentifier=